CLINICAL TRIAL: NCT00506792
Title: A Two-part, Randomized, Double-blind, Placebo-controlled, Ascending Single-dose, Adaptive Study to Evaluate Safety, Tolerability, Pharmacokinetics and Pharmacodynamics of QAU145 Administered Via a Nasal Spray Pump to Patients With Cystic Fibrosis
Brief Title: Safety, Tolerability, Pharmacokinetics, and Pharmacodynamics of QAU145 in Patients With Cystic Fibrosis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CQAU145A2201
Record Dates: First submitted 2007-07-22; First posted 2007-07-25 (Estimated); Last update posted 2020-12-19 (Actual); Status verified 2012-05

CONDITIONS: Cystic Fibrosis
Keywords: Cystic fibrosis, QAU145, nasal potential difference
MeSH Terms: conditions — Cystic Fibrosis

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): QAU145
  Interventions: Drug: QAU145
- 2 (Placebo Comparator): Placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: QAU145
  Arms: 1
Drug: Placebo
  Arms: 2

SUMMARY:
This study will investigate the safety, tolerability, pharmacokinetic, and pharmacodynamic response of patients with cystic fibrosis to administration of QAU145 via intranasal spray.

ELIGIBILITY:
Inclusion Criteria:

* Male and female (women must be post-menopausal or surgically sterile) subjects with cystic fibrosis ages 18 to 50.

Exclusion Criteria:

* Any presence of seasonal or non-seasonal allergies affecting the nose, nasal passages, throat or sinuses within 2 weeks prior to dosing.
* Any upper respiratory tract infection or signs or symptoms within 2 weeks prior to dosing.
* Any presence of nasal polyps or structural abnormalities, frequent history of nose bleeding, or any recent nasal surgery (within 12 weeks prior to dosing).

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 9 (Actual)
Dates: Start 2007-07; Primary Completion 2008-12 (Actual); Study Completion 2009-11 (Actual)

PRIMARY OUTCOMES:
Pharmacodynamic response to single intranasal doses of QAU145 in cystic fibrosis patients using nasal potential difference measurements up to 6 hours post-dose. | Part I: Baseline, 2 hr post dose, after each dose, end of Part I. Part II: Pre dose and 2 hours post each dose

SECONDARY OUTCOMES:
Safety and tolerability of single ascending doses assessed by nasal examinations, adverse events, medications, and a nasal symptom questionnaire. Pharmacokinetics up to 6 hours post-dose | Part I: Throughout study (about 8 weeks) Part II: Throughout study (about 9 weeks)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis, Principal Investigator — Investigative site
Locations (1):
- University of Alabama at Birmingham, Birmingham, Alabama, United States

REFERENCES:
- [Derived] Rowe SM, Reeves G, Hathorne H, Solomon GM, Abbi S, Renard D, Lock R, Zhou P, Danahay H, Clancy JP, Waltz DA. Reduced sodium transport with nasal administration of the prostasin inhibitor camostat in subjects with cystic fibrosis. Chest. 2013 Jul;144(1):200-207. doi: 10.1378/chest.12-2431. PMID 23412700
- See also: Results for CQAU145A2201 from the Novartis Clinical Trials website — https://www.novctrd.com/ctrdweb/trialresult/trialresults/pdf?trialResultId=14397